# Statistical Analysis Plan (SAP)

Study No. NAV3-24

An Evaluation of the Safety of Escalating Doses of Tc 99m Tilmanocept by Intravenous (IV) Injection and a Comparison to Subcutaneous (SC) Injection in Human Immunodeficiency Virus (HIV) Subjects Diagnosed with Kaposi Sarcoma (KS)

Version 1.0

July 23, 2020

Prepared for Navidea Biopharmaceuticals 4995 Bradenton Avenue, Suite 240 Dublin, Ohio 43017

Prepared by
STATKING Clinical Services
759 Wessel Drive
Fairfield, OH 45014
513-858-2989
www.statkingclinical.com



**STATKING Clinical Services** 

## **Approval Page**

By entering into this Statistical Analysis Plan (SAP), the parties acknowledge and agree that this SAP shall be incorporated into and subject to the terms of the Master Services Agreement (MSA). Any changes requested by Client to this SAP shall be subject to Section I.C of the MSA requiring a mutually agreed upon "Change Order" prior to any modification of the procedures set forth herein.

I agree to the format and content of this document.

| And my |
|----------------------------|
| Michael Rosol, PhD |
| Chief Medical Officer |
| Navidea Biopharmaceuticals |

4995 Bradenton Avenue, Suite 240

Dublin, Ohio 43017 mrosol@navidea.com

Approved by:

Approved by:

29 JUL 2020

/29/2020

Bonnie Abbruzzese, MS

Senior Director, Clinical Research and Development

Navidea Biopharmaceuticals

4995 Bradenton Avenue, Suite 240

Dublin, Ohio 43017

babbruzzese@navidea.com

Authored by:

Ian Lees, MS Statistician

STATKING Clinical Services

759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 327

ian@statkingclinical.com

Approved by (internal review):

Lori Christman, PhD

Statistician

STATKING Clinical Services

759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 317

lori@statkingclinical.com

7/30/2020

Clare Geiger, RN Project Manager

STATKING Clinical Services

759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 304

clare@statkingclinical.com

# **Revision History**

N/A

## **Table of Contents**

| 1.0 SYNOPSIS OF STUDY DESIGN PROCEDURES | 7 |
|------------------------------------------------------|----|
| 1.1 Design and Treatment | 7 |
| 1.1.1 Localization Definitions | 8 |
| 1.2 Study Procedures | 8 |
| 1.2.1 Cohorts 1 and 2 | 8 |
| 1.2.2 Cohort 3 | 10 |
| 1.3 Sample Size | 11 |
| 2.0 DATA ANALYSIS CONSIDERATIONS | 12 |
| 2.1 Types of Analyses | 12 |
| 2.2 Analysis Populations | 12 |
| 2.2.1 Subgroup Definitions | 12 |
| 2.3 Missing Data Conventions | 12 |
| 2.4 Interim Analyses | 12 |
| 2.5 Study Center Considerations in the Data Analysis | 13 |
| 2.6 Documentation and Other Considerations | 13 |
| 3.0 ANALYSIS OF BASELINE PATIENT CHARACTERISTICS | 13 |
| 4.0 ANALYSIS OF EFFICACY | 13 |
| 4.1 Description of Efficacy Variables | 13 |
| 4.2 Analysis of Efficacy Variables | 14 |
| 5.0 ANALYSIS OF SAFETY | 16 |
| 6.0 OTHER RELEVANT DATA ANALYSES AND SUMMARIES | 18 |
| 6.1 Subject Completion | 18 |
| 6.2 Study Drug Administration | 18 |

| 6.3 Subject Imaging | 18 |
|---------------------------------------------------------|----|
| 7.0 LIST OF ANALYSIS TABLES, FIGURES AND LISTINGS | 19 |
| 8.0 REFERENCES | 21 |
| APPENDIX A – TABLES, FIGURES AND LISTING SPECIFICATIONS | 22 |
| APPENDIX B – TABLE SHELLS | 24 |

## 1.0 Synopsis of Study Design Procedures

This study will enroll up to fourteen (14) HIV (human immunodeficiency virus) - positive female or male subjects at least 18 years of age who have biopsyconfirmed Kaposi Sarcoma (KS).

The primary objective of this study is:

 To determine the safety of escalating doses of Tc 99m tilmanocept in HIV subjects with biopsy-confirmed KS

The secondary objectives of this study are:

- Concordance between clinical assessment/diagnosis and the localization of Tc 99m tilmanocept by planar and/or SPECT (single photon emission computed tomography) / CT (X-ray computed tomography) imaging in cutaneous and non-cutaneous sites of KS.
- Qualify and quantify Tc 99m tilmanocept localization intensity on imaging with CD206 locale and quantity by histology and immunohistochemistry (IHC) in biopsied KS lesions to determine optimal IV dose.
- Concordance of localization of Tc 99m tilmanocept via IV and SC routes of administration by planar and/or SPECT/CT imaging in cutaneous and non-cutaneous sites of KS.

The exploratory objective of this study is:

 Quantify HHV8 in biopsied KS lesions by real-time polymerase chain reaction (qPCR)

General safety will be evaluated by examining the incidence of adverse events (AEs) and changes over time in laboratory tests, vital signs, ECGs (electrocardiogram) and physical examination findings.

### 1.1 Design and Treatment

This study is a prospective, open-label, single center study of Tc 99m tilmanocept in the localization of KS lesions. Subjects will receive an injection of tilmanocept at one of two mass doses radiolabeled with Tc 99m at one of two radiolabel doses according to the following table:

**Table 1: Description of Cohorts** 

| Cohort Number | Dose | Sample Size |
|---------------|-------------------|-------------|
| 4 | | / |
| 1 | 100μg/5mCi (IV) | 4 |
| 2 | 100μg/10mCi (IV) | 4 |
| 3 | 200μg/5mCi SC, | up to 6 |
| | and 200µg/5mCi IV | |
| | one week later. | |

The 100 or 200  $\mu g$  mass doses will require 1 vial of tilmanocept radiolabeled with the assigned mCi dose delivered in one syringe for IV injections and two syringes for SC injections. Subjects in Cohorts 1 and 2 will have whole body planar imaging beginning 60-75 minutes post-injection followed by optional SPECT/CT of regions of interest. Subjects in Cohort 3 will have a whole-body planar scan with optional SPECT/CT of region of interest scanning beginning at 60- 75 minutes following both the IV and SC injections and 4- 6 hours following SC injection.

#### 1.1.1 Localization Definitions

A localized subject is one for whom Tc 99m tilmanocept by planar and/or SPECT/CT imaging results in the illumination of at least one site relative to background as determined by the nuclear medicine specialist.

A localized KS lesion is a lesion that is both clinically identified or suspected KS (via biopsy-confirmed diagnosis or clinical symptomology) and is illuminated by planar and/or SPECT/CT imaging.

Localization in areas other than KS will also be defined per subject and per area, where these areas are clinically negative KS locations based on clinical symptomology.

## 1.2 Study Procedures

The study includes procedures at screening (within 30 days of injection), preinjection, injection, and post-injection. The post-injection time points include measurements at 30 minutes, 60 - 75 minutes, 4 - 6 hours, and 4 - 10 days postinjection. The following describes the procedures to be conducted on each study day at each time point.

#### 1.2.1 Cohorts 1 and 2

Screening Visit (Visit 1, Day -29 to Day 0): The screening visit will include informed consent, review of study eligibility, allocation of unique subject number, demographic data, medical and surgical history, vital signs (henceforth, vital

signs refers to body temperature, heart rate, systolic and diastolic blood pressure and respiration rate), physical exam including height and body weight, assessment of edema/lymphedema, ECG, blood draw for clinical lab results, cutaneous and non-cutaneous KS evaluation, photographs of all visible cutaneous KS lesions, KS history and classification, urine sample collection for routine urinalysis, urine pregnancy test for women of child-bearing potential, and review of medications.

## Pre-tilmanocept Injection (Visit 2, Day 1):

- Concomitant medication review
- A negative urine pregnancy test for women of child-bearing potential
- Vital signs (within 30 minutes preceding injection)

**Tilmanocept Injection (Day 1):** Based on Cohort assignment, subjects will receive their study drug dose by IV route of administration.

## Post-tilmanocept Injection (Day 1):

- Within 30 minutes post-injection
  - ECG (completed before vital signs)
  - Vital signs
  - Adverse event assessment
- 60- 75 minutes post-injection:
  - Adverse event assessment
  - Whole body planar imaging
  - SPECT/CT imaging of region(s) of interest (optional)
  - After the imaging is complete
    - Blood sample for hematology and serum chemistry
    - Urine sample for routine urinalysis
    - Biopsy of designated non-visceral KS lesion
    - Photograph of biopsy lesion with a measurement scale. This image is to be stored within the subject's research file.

## Follow-Up Telephone Call (7±3 days post-tilmanocept injection):

- Concomitant medication review
- Adverse event assessment

Each subject's participation in the study is complete after the follow-up telephone call.

For determination of secondary endpoints, the Tc 99m tilmanocept whole body planar and SPECT/CT images will be visually assessed for localization by a Nuclear Medicine Physician.

#### 1.2.2 Cohort 3

Screening Visit (Visit 1, Day -29 to Day 0): The screening visit will include informed consent, review of study eligibility, allocation of unique subject number, demographic data, medical and surgical history, vital signs, physical exam including height and body weight, assessment of edema/lymphedema, ECG, blood draw for clinical lab results, cutaneous and non-cutaneous KS evaluation, photographs of all visible cutaneous KS lesions, KS history and classification, urine sample collection for routine urinalysis, urine pregnancy test for women of child-bearing potential, and review of medications.

## Pre-tilmanocept Injection (Visit 2, Day 1):

- Concomitant medication review
- A negative urine pregnancy test for women of child-bearing potential
- Vital signs (within 30 minutes preceding injection)

**Tilmanocept Injection (Day 1):** Subjects will receive their SC study drug dose of 5 mCi Tc 99m/200 μg tilmanocept.

## Post-tilmanocept Injection (Day 1):

- Within 30 minutes post-injection
  - ECG (completed before vital signs)
  - Vital signs
  - Adverse event assessment
- 60- 75 minutes post-injection:
  - o Adverse event assessment
  - Whole body planar imaging
  - SPECT/CT imaging of region(s) of interest (optional)
- 4- 6 hours post-injection:
  - Adverse event assessment
  - Whole body planar imaging
  - SPECT/CT imaging of region(s) of interest (optional)
  - After the imaging is complete
    - Blood sample for hematology and serum chemistry
    - Urine sample for routine urinalysis

### **Pre-tilmanocept Injection (Visit 3, Day 7±3):**

- Concomitant medication review
- A negative urine pregnancy test for women of child-bearing potential
- Vital signs (within 30 minutes preceding injection)

**Tilmanocept Injection (Day 7±3):** Subjects will receive their IV study drug dose of 5 mCi Tc 99m/200 μg tilmanocept.

## Post-tilmanocept Injection (Day 7±3):

- Within 30 minutes post-injection
  - ECG (completed before vital signs)
  - Vital signs
  - Adverse event assessment
- 60- 75 minutes post-injection:
  - Adverse event assessment
  - Whole body planar imaging
  - SPECT/CT imaging of region(s) of interest (optional)
  - o After the imaging is complete
    - Blood sample for hematology and serum chemistry
    - Urine sample for routine urinalysis
    - Biopsy of designated non-visceral KS lesion
    - Photograph of biopsy lesion with a measurement scale. This image is to be stored within the subject's research file.

## Follow-Up Telephone Call (7±3 days post-IV tilmanocept injection):

- Concomitant medication review
- Adverse event assessment

Each subject's participation in the study is complete after the follow-up telephone call.

For determination of secondary endpoints, the Tc 99m tilmanocept whole body planar and SPECT/CT images will be visually assessed for localization by a Nuclear Medicine Physician.

## 1.3 Sample Size

The dose escalation portion of this study is a design with no dose deescalation. The sequential cohort enrollment characteristics of this design do not allow a fixed computation of sample size. In a previous study with subjects receiving a 400 µg dose radiolabeled at 10 mCi (i.e., twice the maximum dose planned for this study), zero (0) subjects had an Adverse Drug Reaction (ADR). Therefore, it is expected that no subjects will have an ADR in this study and that each cohort will enroll the minimum planned sample size of subjects. With 2 cohorts of 4 subjects and one cohort of up to 6 subjects, it is anticipated that the study will enroll no more than n=14 subjects.

## 2.0 Data Analysis Considerations

## 2.1 Types of Analyses

All results will be based on descriptive statistics. Unless otherwise stated, continuous variables will be summarized via sample size, mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized via frequency counts and percentages.

## 2.2 Analysis Populations

The following analysis populations will be defined:

**Safety:** The safety population will include all enrolled subjects who are injected with Tc 99m tilmanocept.

**Intent-to-Diagnose (ITD):** The ITD population will include all subjects who sign informed consent, who are injected with Tc 99m tilmanocept, and who are imaged.

The analysis of all efficacy endpoints will be conducted on the ITD population. The analysis of all safety and baseline subject characteristics will be conducted on the safety population.

## 2.2.1 Subgroup Definitions

Analyses may be performed by dose group (Cohort 1,  $100\mu g/5mCi$ ; Cohort 2,  $100\mu g/10mCi$ ; Cohort 3,  $200\mu g/5mCi$ ) and by route of administration (Cohort 3 SC and IV).

## 2.3 Missing Data Conventions

The analysis of the primary efficacy variables will be carried out on the observed data, i.e., a complete case analysis.

#### 2.4 Interim Analyses

No interim analyses are planned for this study.

## 2.5 Study Center Considerations in the Data Analysis

A study center is defined as a treatment administration site or group of treatment administration sites under the control and supervision of the same Principal Investigator (PI).

Because this is a single-center study, there will be no selective pooling of study centers in the analysis.

#### 2.6 Documentation and Other Considerations

The data analyses will be conducted using SAS© Software, version 9.4 or later.

## 3.0 Analysis of Baseline Patient Characteristics

Baseline and demographic characteristics will be summarized by dose group for all subjects in the safety population. Continuous variables will be displayed via summary statistics (mean, median, sample size, standard deviation, minimum, and maximum). Categorical variables will be summarized via counts and percentages.

A detailed listing of demographic data for each subject will also be provided as shown in Appendix B.

## 4.0 Analysis of Efficacy

## 4.1 Description of Efficacy Variables

Secondary objectives of the study are to determine the concordance between clinical assessment/diagnosis and the localization of Tc 99m tilmanocept by planar and/or SPECT/CT imaging in cutaneous and non-cutaneous sites of KS; to qualify and quantify Tc 99m tilmanocept localization intensity on imaging with CD 206 locale and quantity by histology and IHC in biopsied KS lesions to determine the optimal IV dose; and concordance of localization of Tc 99m tilmanocept via IV and SC routes of administration by planar and/or SPECT/CT imaging in cutaneous and non-cutaneous sites of KS. The relevant endpoints are the following:

- Per subject localization rate of Tc 99m tilmanocept in at least one KS suspected or confirmed lesion by planar and/or SPECT/CT imaging
- Per lesion/region concordance of Tc 99m localization with anatomical areas of active KS defined by confirmed diagnosis or clinical symptomology

- Localization intensity for each biopsied and clinically defined lesion localized on imaging following IV injection as determined by quantitative SPECT gamma counts
- Per biopsied lesion proportion of CD206-expressing cells and proportion of HHV8-expressing cells as determined by histology and relative IHC fluorescence
- Per lesion/region concordance of IV vs SC Tc 99m localization with anatomical areas of active KS defined by confirmed diagnosis or clinical symptomology.
- Per subject localization rate of Tc 99m tilmanocept in areas other than KS by planar and/or SPECT/CT imaging
- Per area localization rate of Tc 99m tilmanocept in the most frequently identified areas other than KS by planar and/or SPECT/CT imaging

An exploratory objective of the study is to use quantitative Polymerase Chain Reaction (qPCR) methods to measure the amount of Human Herpes Virus 8 (HHV8) present in the biopsy tissue.

The relevant variables are the following:

- Nuclear medicine specialist determination of presence/absence of illumination (i.e., localization positive or negative per anatomic site) relative to background from planar and/or SPECT/CT imaging results for each subject;
- Clinically identified presence or absence of KS based on any previous diagnostic evaluation;
- Proportion of CD206-expressing cells (IHC fluorescence);
- Quantitative SPECT gamma counts for each biopsied lesion localized on imaging following IV injection; and,
- HHV8 concentrations as determined by gPCR for each biopsied lesion.

The calculations and analyses pertaining to each of the variables are shown in Sections 4.2.

## 4.2 Analysis of Efficacy Variables

#### **Localization in KS Sites**

The number and percentage of subjects with at least one biopsy-confirmed or clinically suspected KS lesion that has localized with Tc 99m tilmanocept by planar and/or SPECT/CT imaging will be computed. A 95% exact confidence interval on the per-subject localization rate will be computed. This analysis will be performed by dose group and route of administration.

Per-lesion/region localization of Tc 99m tilmanocept by planar and/or SPECT/CT imaging will be computed across all biopsy-confirmed or clinically suspected KS lesions of all subjects. A 95% exact confidence interval on the per-lesion/region localization will be calculated. This analysis will be performed by dose group and route of administration.

An analysis table will also be provided to display the counts of KS lesions localized by imaging that were not previously identified clinically.

Concordance between IV and SC tilmanocept in biopsy-confirmed or clinically-suspected KS lesion sites will be assessed with a cross-tabulation of the IV and SC findings, including the joint probability distribution. The sampling unit for this analysis will be the site. An exact conditional version of McNemar's test will be performed to test the hypotheses

$$H_0: \pi_{IV} = \pi_{SC}$$
  
 $H_A: \pi_{IV} \neq \pi_{SC}$ ,

where  $\pi_{IV}$  and  $\pi_{SC}$  represent the probabilities of localization with IV (only) tilmanocept and SC (only) tilmanocept, respectively. In addition, the number and proportion of subjects with concordance and reverse concordance of observed sites of discrete localization of Tc 99m tilmanocept following IV and SC localization will be summarized.

## Localization Intensity by Planar and/or SPECT/CT Imaging

Tc 99m tilmanocept average pixel intensity and percent above background will be summarized with descriptive statistics (mean, standard deviation, minimum, median, maximum, and range) for each biopsied lesion localized on imaging following IV injection of Tc 99m tilmanocept by dose group. Summary statistics will be presented separately by imaging type (planar, SPECT/CT).

## **Proportion of CD206-expressing Cells**

Per biopsied-lesion proportion of CD206-expressing cells as determined by histology and IHC fluorescence will be summarized by descriptive statistics (mean, standard deviation, minimum, median, maximum, and range) by dose group.

#### **Localization in Non-KS Sites**

The number and percentage of subjects with at least one anatomical site other than KS that has been localized with Tc 99m tilmanocept by planar and/or SPECT/CT imaging will be computed. A 95% exact confidence interval on the per subject localization rate will be computed. This analysis will be performed by dose group and route of administration.

Locations showing localization of Tc 99m tilmanocept by planar and/or SPECT/CT imaging will be computed across all sites other than biopsyconfirmed or clinically suspected KS sites of all subjects. A 95% exact confidence interval on per location localization will be calculated. (i.e. the rate of localization of each site with respect to the number of subjects). This analysis will be performed by dose group and route of administration.

## 5.0 Analysis of Safety

Adverse Drug Reactions (ADRs) are defined as all noxious and unintended responses to a medicinal product related to any dose or dose regimen. The phrase 'responses to a medicinal product' means that a causal relationship between a medicinal product and an adverse event. The primary safety variable is the proportion of patients experiencing at least one ADR. The number and percentage of subjects with ADRs will be tabulated by dose group and overall. Other safety endpoints are noted below.

## **Analysis of Safety Endpoints**

Attention shall be paid to the occurrence of adverse events (AEs) from the time of signing informed consent until exit from the study. Events occurring prior to Tc 99m tilmanocept administration will be recorded in the subject's medical history unless determined to be related to the study procedure. A treatment emergent adverse event (TEAE) is defined as an adverse event whose start date is on or after the first study drug administration date. If the study drug administration date and/or the AE start date are missing, the AE will be considered treatment emergent.

Prior to analysis, all AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The MedDRA version used will be stated in the final validated tables. Based on these coded terms, AEs and TEAEs will be summarized by dose group and overall as follows:

- by system organ class and preferred terms;
- by system organ class and preferred terms and relation to study drug; and,
- by system organ class and preferred terms and severity.

In addition to the above endpoints, the following describes the analyses of the other safety data being collected for the study.

#### **Vital Signs**

Vital signs will include heart rate, blood pressure, respiration rate, and body temperature. Vital signs will be taken during screening, prior to study drug administration on Day 1 (and Day 7 [± 3] for Cohort 3), and within 30 minutes following study drug administration. For each vital sign, summary statistics

(mean, standard deviation, minimum, median, maximum, range, n) on the raw values as well as their changes from pre-injection on Day 1 (and Day 7 [± 3] for Cohort 3) will be presented by dose group and overall. Time points included in this analysis are Day 1 (and Day 7 [± 3] for Cohort 3) within 30 minutes pre-injection and within 30 minutes post-Injection. If repeat vital signs are taken at a given time point, then the last measurement will be used for the analysis tables. A shift table will be created showing shifts Abnormal/Abnormal, Abnormal/Normal, Normal/Normal, Normal/Normal from pre-injection to post-injection of Tc 99m tilmanocept. This analysis will be performed by dose group and overall.

All vital signs will be listed, including those not presented in the analysis tables.

## **Physical Exams**

A complete physical exam will be performed during screening. A data listing of the physical exam results will be created as shown in Appendix B.

#### **Concomitant Medications**

All concomitant medications will be coded with WHO Drug Dictionary (Uppsala Monitoring Centre) version March 2017 or later. A data listing will be constructed with Preferred Term, Verbatim Term, ATC Level 1 Code, and ATC Level 4 Code. A summary table will be provided to show the counts and percentages of subjects taken medications by ATC Level 4 Code and Preferred Term by dose group and overall.

#### **Clinical Laboratory Parameters**

Changes in hematology, clinical serum chemistry and urinalysis between screening (i.e., baseline) and the post-injection time point will be calculated, and descriptive statistics will be calculated on the raw and change from baseline values by dose group and overall. A copy of the normal laboratory values for all laboratories utilized for this study will be submitted to the Sponsor (or designee) prior to initiation of the study. A shift table will be created showing shifts Abnormal/Abnormal, Abnormal/Normal, Normal/Normal, Normal/Normal from screening baseline to post-injection of Tc 99m tilmanocept. This analysis will be performed by dose group and overall.

#### **ECG**

ECG recordings will be obtained during screening (i.e., baseline) and within 30 minutes following study drug administration. ECG parameters (heart rate, PR interval, QRS interval, QT interval, and QTcF interval) will be summarized as raw values and change-from-baseline (CFB). A shift table will be created showing shifts Abnormal/Abnormal, Abnormal/Normal, Normal/Abnormal, Normal/Normal from screening baseline to post-injection of Tc 99m tilmanocept. Both the quantitative and shift table analyses will be performed by dose group and overall.

## 6.0 Other Relevant Data Analyses and Summaries

## 6.1 Subject Completion

A table will be constructed with counts of screen failures and enrolled subjects. Of those enrolled, counts and percentages of the number of subjects withdrawing from the study before study completion and the number completing the study will be displayed. For those subjects that withdraw before completion of the study, counts and percentages of the reasons for withdrawal will be tabulated. The table will include summary counts and percentages by dose group and overall. A data listing of all subject completion and withdrawal data will also be constructed.

## **6.2 Study Drug Administration**

The mass dose and radioactivity of Tc 99m tilmanocept injected will be summarized by dose group and overall.

## 6.3 Subject Imaging

Each subject will undergo whole body planar imaging. SPECT/CT imaging of region(s) of interest is optional for each subject. Results of all imaging procedures will be listed.

# 7.0 List of Analysis Tables, Figures and Listings

| Table<br>No. | Table Title | Included<br>in Final<br>Tables | Shown in Appendix B |
|---|---|---|---|
| 1 | Subject Disposition by Cohort | X | X |
| 2 | Demographics and Baseline Data Summary Statistics by Cohort – Continuous Variables (Safety Population) | X | X |
| 3 | Demographics and Baseline Data Summary Statistics<br>by Cohort – Categorical Variables (Safety Population) | Х | Х |
| 4 | Summary of Study Drug Administration by Cohort (Safety Population) | Х | Х |
| 5 | Subject-Level Localization of KS Lesions – Nuclear Medicine Findings (ITD Population) | Х | Х |
| 6 | Lesion-Level Localization of KS Lesions – Nuclear Medicine Findings (ITD Population) | Х | Х |
| 7 | Additional KS Lesions Identified from Imaging That<br>Were Not Seen Clinically – Nuclear Medicine Findings<br>(ITD Population) | х | Х |
| 8 | Lesion-Level Non-Localization of KS Lesions – Nuclear Medicine Findings (ITD Population) | Х | Х |
| 9 | Number and Percentage of Concordant and Reverse Concordant Lesions (ITD Population) | Х | Х |
| 10 | Summary of Imaging-Localized Biopsied Lesion Localization Intensity by Cohort – Imaging = Planar (ITD Population) | Х | X |
| 11 | Summary of Imaging-Localized Biopsied Lesion Localization Intensity by Cohort – Imaging = SPECT/CT (ITD Population) | х | Х |
| 12 | Summary of Per Biopsied Lesion Proportion of CD206-<br>Expressing Cells and Proportion of HHV8-Expressing<br>Cells by IHC (ITD Population) | Х | Х |
| 13 | Summary of Per Biopsied Lesion HHV8 Quantitation by qPCR (ITD Population) | Х | Х |
| 14 | Subject-Level Localization in Areas Other Than KS Sites – Nuclear Medicine Findings (ITD Population) | Х | Х |
| 15 | Site-Level Localization in Areas Other Than KS Sites – Nuclear Medicine Findings (ITD Population) | Х | Х |
| 16 | Number and Percent of Subjects with Adverse Events (Safety Population) | Х | Х |
| 17 | Summary of Adverse Events (Safety Population) | X | X |
| 18 | Number and Percent of Subjects with Treatment<br>Emergent Adverse Events (Safety Population) | Х | Х |
| 19 | Summary of Treatment Emergent Adverse Events (Safety Population) | Х | Х |
| 20 | Number and Percent of Subjects with Adverse Drug Reactions (Safety Population) | Х | Х |
| 21 | Number and Percent of Subjects with Serious Adverse Events (Safety Population) | Х | Х |
| 22 | Vital Sign Parameters Summary Statistics (Safety Population) | Х | Х |

| Table<br>No. | Table Title | Included<br>in Final<br>Tables | Shown in<br>Appendix B |
|---|---|---|---|
| 23 | Vital Sign Shift Table (Safety Population) | X | X |
| 24 | Clinical Laboratory Parameters Summary Statistics (Safety Population) | X | X |
| 25 | Clinical Laboratory Parameters Shift Table (Safety Population) | Х | Х |
| 26 | Electrocardiogram Parameters Summary Statistics (Safety Population) | Х | Х |
| 27 | Electrocardiogram Shift Table (Safety Population) | Х | X |
| 28 | Number and Percent of Subjects Taking Concomitant Medications (Safety Population) | Х | Х |

| Listing<br>No. | Data Listing Title | Included<br>in Final<br>Listings | Shown in Appendix B |
|---|---|---|---|
| NO. | Data Listing Title | Listings | Appelluix B |
| DL1 | Subject Disposition Data Listing | X | Х |
| DL2 | Inclusion/Exclusion Data Listing | X | X |
| DL3 | Protocol Deviations Data Listing | Х | X |
| DL4 | Demographics Data Listing | X | X |
| DL5 | Subjects Excluded from ITD Population Data Listing | X | X |
| DL6 | Medical History Data Listing | X | X |
| DL7 | Prior and Concomitant Medications Data Listing | X | X |
| DL8 | Adverse Events Data Listing | X | X |
| DL9 | Subject Laboratory Profiles - Hematology Data Listing | X | X |
| DL10 | Subject Laboratory Profiles – Serum Chemistry Data Listing | X | X |
| DL11 | Subject Laboratory Profiles – Urinalysis Data Listing | Х | Х |
| DL12 | Electrocardiogram Data Listing | X | Х |
| DL13 | Physical Exam Data Listing | X | X |
| DL14 | Vital Signs Data Listing | X | X |
| DL15 | Study Drug Administration Data Listing | X | X |
| DL16 | Post-Injection Imaging Data Listing | X | X |
| DL17 | Quantitative Imaging Results Data Listing | X | X |
| DL18 | Qualitative Imaging Results Data Listing | X | X |
| DL19 | Lesion Biopsy Results Data Listing | X | X |
| DL20 | Clinical KS Lesion Assessment Listing | X | X |
| DL21 | Telephone Follow Up Contact Data Listing | X | X |

## 8.0 References

NA

## Appendix A – Tables, Figures and Listing Specifications

#### Orientation

Tables, figures, and listings will be displayed in landscape.

## **Margins**

Margins will be 1 inch on all sides. Table, figure, and listing boundaries will not extend into the margins.

#### **Font**

Courier New, 8 point.

#### Headers

The table number will be on the second line of the title area. The title area will contain the Sponsor name, the study number, and the name of the table. The title area will contain the page number (Page x of y) on the far right, one line above the name of the table.

#### **Footers**

- The first line will be a solid line.
- Next will be any footnotes regarding information displayed in the table.
- Below these footnotes will be displayed "STATKING Clinical Services (Date)" on the far left.
- The last line will display the name of the SAS program that generated the table and (if applicable) the source data reference.

### **Table Disclaimer**

The format of the mock tables shown in the appendix of this Statistical Analysis Plan (SAP) will be the format of the deliverable tables to the extent that Word document constructed tables can match production tables produced by SAS. This formatting includes the content and format of the header and footer areas of the tables. The Sponsor agrees to the format of the tables as shown in the appendix.

Further programming charges will be applicable for changes in the format of tables (including title statements, notes, data dependent footnotes, etc.) made after the approval of the SAP.

## **Missing Values**

All missing values will be displayed on the output tables/listings as blanks.

## **Computation Values for Study Dates**

The date format to be used is dd-mmm-yyyy. Missing parts of dates are not shown (e.g., for a missing day value, the value displayed is in mmm-yyyy format). When date computations are necessary, the following table indicates the substitutions used in order to make those computations.

| Scenario | Value Used for Computations |
|---|---|
| Start date – Missing month and day values | January 1 of the indicated year |
| Start date – Missing day values | The first day of the indicated month |
| Stop date – Missing month and day values | December 31 of the indicated year |
| Stop date – Missing day values | The last day of the indicated month |

Appendix B – Table Shells

Page x of y

Table 1. Subject Disposition by Cohort Navidea Biopharmaceuticals - Study No. NAV3-24

| | | Сс | hort 1 | Со | hort 2 | Со | hort 3 | ΟV | verall |
|---|---|---|---|---|---|---|---|---|---|
| Screen Failures | | | XX | | XX | | XX | | XX |
| Enrolled | | | xx | | xx | | xx | | xx |
| Completed | | XX | (xxx%) | xx | (xxx%) | xx | (xxx%) | XX | (xxx%) |
| Withdrawn | | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| Reason for Withdrawal | Adverse Event | XX | (xxx%) | xx | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| | Lost To Follow-Up | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| | Death | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| | Physician Decision | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| | Protocol Deviation | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| | Study Terminated by | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| | Sponsor | | | | | | | | |
| | Withdrawal by Subject | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| | Other | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |

The denominator for all percentages in the table is the number of enrolled subjects in the respective cohort and overall. Cohort  $1 = 100\mu g/5mCi$  IV; Cohort  $2 = 100\mu g/10mCi$  IV; Cohort  $3 = 200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 2. Demographics and Baseline Data Summary Statistics by Cohort - Continuous Variables
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

| | Group | | | | | | |
|---|---|---|---|---|---|---|---|
| Variable | | Mean | Std Dev | n | Min | Max | Median |
| Age (years) | Cohort 1 | XXX | XXX | XXX | XXX | XXX | XXX |
| | Cohort 2 | XXX | XXX | XXX | XXX | XXX | XXX |
| | Cohort 3 | XXX | XXX | XXX | XXX | XXX | XXX |
| | Overall | XXX | xxx | XXX | XXX | XXX | XXX |
| Height (in) | Cohort 1 | XXX | xxx | XXX | xxx | xxx | xxx |
| , , , | Cohort 2 | xxx | XXX | XXX | xxx | xxx | xxx |
| | Cohort 3 | xxx | XXX | XXX | xxx | xxx | XXX |
| | Overall | XXX | XXX | XXX | XXX | XXX | xxx |
| Weight (lb) | Cohort 1 | XXX | xxx | XXX | xxx | XXX | xxx |
| | Cohort 2 | xxx | XXX | xxx | xxx | xxx | xxx |
| | Cohort 3 | xxx | xxx | XXX | xxx | xxx | XXX |
| | Overall | XXX | xxx | XXX | XXX | XXX | XXX |
| Number of KS lesions <sup>a</sup> | Cohort 1 | XXX | xxx | XXX | xxx | XXX | xxx |
| | Cohort 2 | XXX | XXX | xxx | xxx | xxx | xxx |
| | Cohort 3 | xxx | XXX | xxx | XXX | xxx | xxx |
| | Overall | XXX | XXX | XXX | XXX | XXX | XXX |

 $<sup>^{</sup>a}$  Number of KS lesions identified in screening, including cutaneous and non-cutaneous lesions. Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC.

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 3. Demographics and Baseline Data Summary Statistics by Cohort - Categorical Variables
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

| Demographics<br>Variable | Category | Cohort 1 (N=xxx) | Cohort 2 (N=xxx) | Cohort 3 (N=xxx) | Overall (N=xxx) |
|---|---|---|---|---|---|
| Gender | Male | XXX | XXX | XXX | XXX |
| | | (xxx%) | (xxx%) | (xxx%) | (xxx%) |
| | Female | XXX | XXX | XXX | XXX |
| | | (xxx%) | (xxx%) | (xxx%) | (xxx%) |
| Race | American Indian or Alaska | XXX | xxx | xxx | xxx |
| | Native | (xxx%) | (xxx%) | (xxx%) | (xxx%) |
| | Asian | XXX | XXX | XXX | XXX |
| | | (xxx%) | (xxx%) | (xxx%) | (xxx%) |
| | Black or African American | XXX | XXX | XXX | XXX |
| | | (xxx%) | (xxx%) | (xxx%) | (xxx%) |
| | Native Hawaiian or Other | XXX | XXX | XXX | XXX |
| | Pacific Islander | (xxx%) | (xxx%) | (xxx%) | (xxx%) |
| | White | XXX | XXX | XXX | XXX |
| | | (xxx%) | (xxx%) | (xxx%) | (xxx%) |
| | Other | XXX | XXX | XXX | XXX |
| | | (xxx%) | (xxx%) | (xxx%) | (xxx%) |
| Ethnicity | Hispanic or Latino | xxx | xxx | xxx | xxx |
| - | - | (xxx%) | (xxx%) | (xxx%) | (xxx%) |
| | Not Hispanic or Latino | xxx | xxx | xxx | xxx |
| | - | (xxx%) | (xxx%) | (xxx%) | (xxx%) |
| | | | | | , |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 4. Summary of Study Drug Administration by Cohort Navidea Biopharmaceuticals - Study No. NAV3-24 Safety Population (N=xxx)

| | Group | Mean | Std Dev | n | Min | Max | Median |
|-------------------|-------------|------|---------|----|------|------|--------|
| Tc 99m Dose (mCi) | Cohort 1 IV | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| | Cohort 2 IV | xxxx | XXXX | XX | XXXX | XXXX | XXXX |
| | Cohort 3 IV | xxxx | XXXX | XX | XXXX | XXXX | XXXX |
| | Cohort 3 SC | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| Mass Dose (µg) | Cohort 1 IV | xxxx | xxxx | XX | xxxx | xxxx | xxxx |
| | Cohort 2 IV | xxxx | XXXX | XX | XXXX | XXXX | XXXX |
| | Cohort 3 IV | xxxx | XXXX | XX | XXXX | XXXX | XXXX |
| | Cohort 3 SC | xxxx | XXXX | xx | XXXX | XXXX | XXXX |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC.

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 5. Subject-Level Localization of KS Lesions-Nuclear Medicine Findings
Navidea Biopharmaceuticals - Study No. NAV3-24

ITD Population (N=xxx)

| _Group | Number<br>of Subjects | Number<br>(Proportion)<br>Localized | 95% Exact One-<br>Sided Binomial<br>CI for<br>Proportion |
|---|---|---|---|
| Cohort 1 IV | xx | xxx (xxx) | (xxx, xxx) |
| Cohort 2 IV | xx | xxx (xxx) | (xxx, xxx) |
| Cohort 3 IV | XX | xxx (xxx) | (xxx, xxx) |
| Cohort 3 SC | XX | xxx (xxx) | (xxx, xxx) |
| All Cohorts<br>Combined | xx | xxx (xxx) | (xxx, xxx) |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 6. Lesion-Level Localization of KS Lesions-Nuclear Medicine Findings
Navidea Biopharmaceuticals - Study No. NAV3-24
ITD Population (N=xxx)

| Group | Number of<br>Clinically<br>Identified<br>Lesions <sup>a</sup> | Number<br>(Proportion)<br>Localized by<br>Imaging | 95% Exact One-<br>Sided Binomial<br>CI for<br>Proportion |
|---|---|---|---|
| Cohort 1 IV | xx | xxx (xxx) | (xxx, xxx) |
| Cohort 2 IV | xx | xxx (xxx) | (xxx, xxx) |
| Cohort 3 IV | xx | xxx (xxx) | (xxx, xxx) |
| Cohort 3 SC | xx | xxx (xxx) | (xxx, xxx) |
| All Cohorts<br>Combined | xx | xxx (xxx) | (xxx, xxx) |

 $<sup>^{\</sup>rm a}$  Number of cutaneous and non-cutaneous lesions identified in screening. Cohort 1 = 100µg/5mCi IV; Cohort 2 = 100µg/10mCi IV; Cohort 3 = 200µg/5mCi IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 7. Additional KS Lesions Identified from Imaging That Were Not Seen Clinically - Nuclear

Medicine Findings

Navidea Biopharmaceuticals - Study No. NAV3-24

ITD Population (N=xxx)

| Group | Number of<br>Identified<br>Lesions | Number (Proportion) of<br>Subjects with at Least<br>1 Identified Lesion |
|---|---|---|
| Cohort 1 IV | XX | xxx (xxx) |
| Cohort 2 IV | xx | xxx (xxx) |
| Cohort 3 IV | xx | xxx (xxx) |
| Cohort 3 SC | xx | xxx (xxx) |
| All Cohorts<br>Combined | xx | xxx (xxx) |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 8. Lesion-level Non-Localization of KS Lesions - Nuclear Medicine Findings
Navidea Biopharmaceuticals - Study No. NAV3-24

ITD Population (N=xxx)

| Group | Number of<br>Clinically<br>Identified<br>Lesions <sup>a</sup> | Number<br>(Proportion) Not<br>Localized by<br>Imaging | 95% Exact One-<br>Sided Binomial<br>CI for<br>Proportion |
|---|---|---|---|
| Cohort 1 IV | XX | xxx (xxx) | (xxx, xxx) |
| Cohort 2 IV | XX | xxx (xxx) | (xxx, xxx) |
| Cohort 3 IV | XX | xxx (xxx) | (xxx, xxx) |
| Cohort 3 SC | XX | xxx (xxx) | (xxx, xxx) |
| All Cohorts<br>Combined | xx | xxx (xxx) | (xxx, xxx) |

 $<sup>^{\</sup>rm a}$  Number of cutaneous and non-cutaneous lesions identified in screening. Cohort 1 = 100µg/5mCi IV; Cohort 2 = 100µg/10mCi IV; Cohort 3 = 200µg/5mCi IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 9. Number and Percentage of Concordant and Reverse Concordant Lesions Navidea Biopharmaceuticals - Study No. NAV3-24 ITD Population (N=xxx)

| | SC | Result | | | | |
|---|---|---|---|---|---|---|
| IV Result | Localized | Not Localized | <br>Total | Concordance | Reverse<br>Concordance | p-Value<br>(McNemar's Test) |
| Localized | xx (xxx%) | xx(xxx%) | xx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx |
| Not Localized | xx(xxx%) | xx(xxx%) | xx(xxx%) | | | |
| Total | xx(xxx%) | xx (xxx%) | | | | |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Page x of y

Table 10. Summary of Imaging-Localized Biopsied Lesion Localization Intensity by Cohort - Imaging = Planar

Navidea Biopharmaceuticals - Study No. NAV3-24

ITD Population (N=xxx)

| | | | Std | | | | |
|---|---|---|---|---|---|---|---|
| Group | Variable <sup>a</sup> | Mean | Dev | n | Min | Max | Median |
| Cohort 2 IV | Avg Pixel Intensity | xx | xx | XX | XX | XX | xx |
| | Percent Above Background | XX | XX | XX | XX | XX | XX |
| Cohort 3 IV | Avg Pixel Intensity | xx | XX | xx | XX | xx | XX |
| | Percent Above Background | XX | XX | XX | XX | XX | XX |
| All Cohorts Combined | Avg Pixel Intensity | XX | XX | XX | XX | XX | XX |
| | Percent Above Background | XX | XX | XX | XX | XX | XX |

 $<sup>^{\</sup>rm a}$  All summary statistics are performed on the subject level. Cohort 1 = 100µg/5mCi IV; Cohort 2 = 100µg/10mCi IV; Cohort 3 = 200µg/5mCi IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 11. Summary of Imaging-Localized Biopsied Lesion Localization Intensity by Cohort - Imaging = SPECT/CT

Navidea Biopharmaceuticals - Study No. NAV3-24

ITD Population (N=xxx)

| | | | Std | | | | |
|---|---|---|---|---|---|---|---|
| Group | Variable <sup>a</sup> | Mean | Dev | n | Min | Max | Median |
| Cohort 2 IV | Avg Pixel Intensity | xx | xx | XX | XX | XX | XX |
| | Percent Above Background | XX | XX | XX | XX | XX | XX |
| Cohort 3 IV | Avg Pixel Intensity | xx | XX | XX | XX | XX | XX |
| | Percent Above Background | XX | XX | XX | XX | XX | XX |
| All Cohorts Combined | Avg Pixel Intensity | XX | XX | XX | XX | XX | XX |
| | Percent Above Background | XX | XX | XX | XX | XX | XX |

 $<sup>^{\</sup>rm a}$  All summary statistics are performed on the subject level. Cohort 1 = 100µg/5mCi IV; Cohort 2 = 100µg/10mCi IV; Cohort 3 = 200µg/5mCi IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 12. Summary of Per Biopsied Lesion Proportion of CD206-Expressing Cells and Proportion of HHV8-Expressing Cells by IHC

Navidea Biopharmaceuticals - Study No. NAV3-24

ITD Population (N=xxx)

| Group | Variable | Mean | Std<br>Dev | n | Min | Max | Median |
|---|---|---|---|---|---|---|---|
| Cohort 2 | Proportion of CD206-Expressing Cells | XX | xx | XX | XX | XX | XX |
| | Proportion of HHV8-Expressing Cells | XX | XX | XX | XX | XX | XX |
| Cohort 3 | Proportion of CD206-Expressing Cells | XX | xx | XX | XX | XX | XX |
| | Proportion of HHV8-Expressing Cells | XX | XX | XX | XX | XX | XX |
| All Cohorts | Proportion of CD206-Expressing Cells | xx | xx | xx | xx | XX | XX |
| | Proportion of HHV8-Expressing Cells | XX | xx | XX | XX | XX | XX |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC.

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas
Page x of y

Table 13. Summary of Per Biopsied Lesion HHV8 Quantitation by qPCR
Navidea Biopharmaceuticals - Study No. NAV3-24
ITD Population (N=xxx)

| Group | Variable (Unit) | Mean | Std<br>Dev | n | Min | Max | Median |
|----------|-----------------|------|------------|----|-----|-----|--------|
| Cohort 2 | HHV8 (RFU) | XX | XX | XX | XX | xx | XX |
| Cohort 3 | HHV8 (RFU) | XX | xx | XX | XX | XX | XX |

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Table 14. Subject-Level Localization in Areas Other Than KS Sites - Nuclear Medicine Findings
Navidea Biopharmaceuticals - Study No. NAV3-24

ITD Population (N=xxx)

| Group | Number of<br>Subjects | Number<br>(Proportion)<br>Localized | 95% Exact One-<br>Sided Binomial<br>CI for<br>Proportion |
|---|---|---|---|
| Cohort 1 IV | xx | xxx (xxx) | (xxx, xxx) |
| Cohort 2 IV | XX | xxx (xxx) | (xxx, xxx) |
| Cohort 3 IV | xx | xxx (xxx) | (xxx, xxx) |
| Cohort 3 SC | xx | xxx (xxx) | (xxx, xxx) |
| All Cohorts Combined | xx | xxx (xxx) | (xxx, xxx) |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC.

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 15. Site-Level Localization in Areas Other Than KS Sites - Nuclear Medicine Findings
Navidea Biopharmaceuticals - Study No. NAV3-24

ITD Population (N=xxx)

| | | Number<br>(Proportion) of | 95% Exact One-<br>Sided Binomial |
|---|---|---|---|
| | | Subjects with Site | CI for |
| Group | Anatomical Site | Localized | Proportion |
| | | | _ |
| Cohort 1 IV | xxxxxxxxxxxxxx | xxx (xxx) | (xxx, xxx) |
| | xxxxxxxxxxxxxx | | |
| Cohort 2 IV | xxxxxxxxxxxxxx | xxx (xxx) | (xxx, xxx) |
| | xxxxxxxxxxxxxx | | |
| Cohort 3 IV | xxxxxxxxxxxxxx | xxx (xxx) | (xxx, xxx) |
| | xxxxxxxxxxxxxx | | |
| Cohort 3 SC | xxxxxxxxxxxxxx | xxx (xxx) | (xxx, xxx) |
| | xxxxxxxxxxxxxx | | |
| All Cohorts Combined | xxxxxxxxxxxxxx | xxx (xxx) | (xxx, xxx) |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 16. Number and Percent of Subjects with Adverse Events
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

| Adverse Event Categorya: | Cohort 1 (N=xxx) | Cohort 2 (N=xxx) | Cohort 3 (N=xxx) | Overall (N=xxx) |
|---|---|---|---|---|
| Total Number of Adverse Events | xxx xxx | | xxx | xxx |
| Subjects with at Least One Adverse Event | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX.
Cohort 1 = 100μg/5mCi IV; Cohort 2 = 100μg/10mCi IV; Cohort 3 = 200μg/5mCi IV and SC.
STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxxx.sas

Page x of y

Table 17. Summary of Adverse Events Navidea Biopharmaceuticals - Study No. NAV3-24 Safety Population (N=xxxx)

| | Cohort 1<br>(N=xxx) | Cohort 2 (N=xxx) | Cohort 3 (N=xxx) | Overall (N=xxx) |
|---|---|---|---|---|
| Subjects with at Least One<br>Adverse Event | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Maximum AE Severity Grade | | | | |
| Mild | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Moderate | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Severe | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Highest Relationship of AE to Tc 99m Tilmanocept | | | | |
| Definitely Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Possibly [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Definitely [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Highest Relationship of AE to Study Procedure | | | | |
| Definitely Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Possibly [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Definitely [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Subjects with at Least One<br>Serious Adverse Event | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC.

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 18. Number and Percent of Subjects with Treatment Emergent Adverse Events
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

| Adverse Event Categorya: | Cohort 1<br>(N=xxx) | Cohort 2 (N=xxx) | Cohort 3 (N=xxx) | Overall<br>(N=xxx) |
|---|---|---|---|---|
| Total Number of Treatment Emergent Adverse Events (TEAEs) | xxx | xxx | xxx | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) |

 $<sup>^{\</sup>rm a}$  Adverse events coded with MedDRA Coding Dictionary Version XXX. Cohort 1 = 100µg/5mCi IV; Cohort 2 = 100µg/10mCi IV; Cohort 3 = 200µg/5mCi IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxxx.sas

Page x of y

Table 19. Summary of Treatment Emergent Adverse Events
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxxx)

| | Cohort 1<br>(N=xxx) | Cohort 2<br>(N=xxx) | Cohort 3<br>(N=xxx) | Overall (N=xxx) |
|---|---|---|---|---|
| Subjects with at Least One<br>Treatment Emergent Adverse<br>Event (TEAE) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Maximum TEAE Severity Grade | | | | |
| Mild | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Moderate | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Severe | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Highest Relationship of TEAE to Tc 99m Tilmanocept | | | | |
| Definitely Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Possibly [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Definitely [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Highest Relationship of TEAE to Study Procedure | | | | |
| Definitely Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Possibly [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Definitely [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Subjects with at Least One<br>Serious TEAE Adverse Event | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC.

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 20. Number and Percent of Subjects with Adverse Drug Reactions
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

| Adverse Event Categorya: | Cohort 1 (N=xxx) | Cohort 2<br>(N=xxx) | Cohort 3<br>(N=xxx) | Overall<br>(N=xxx) |
|---|---|---|---|---|
| Total Number of Adverse Drug Reactions <sup>b</sup> | xxx | xxx | xxx | xxx |
| Subjects with at Least One Adverse Drug Reaction | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 Preferred Term 1 | xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC.

STATKING Clinical Services (DD-MMM-YYYY)

a Adverse events coded with MedDRA Coding Dictionary Version XXX.

b Adverse drug reactions are defined as all noxious and unintended responses to a medicinal product related to any dose or dose regimen. The phrase 'responses to a medicinal product' means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility, i.e. the relationship cannot be ruled out.

Page x of y

Table 21. Number and Percent of Subjects with Serious Adverse Events Navidea Biopharmaceuticals - Study No. NAV3-24 Safety Population (N=xxx)

| Adverse Event Categorya: | Cohort 1<br>(N=xxx) | Cohort 2<br>(N=xxx) | Cohort 3 (N=xxx) | Overall<br>(N=xxx) |
|---|---|---|---|---|
| Total Number of Serious Adverse<br>Events | xxx | xxx | xxx | xxx |
| Subjects with at Least One<br>Serious Adverse Event | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%) xxx (xxx%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | xxx (xxx%) xxx (xxx%) xxx (xxx%) | xxx (xxx%) xxx (xxx%) | xxx (xxx%) xxx (xxx%) xxx (xxx%) | xxx (xxx%) xxx (xxx%) xxx (xxx%) |

a Adverse events coded with MedDRA Coding Dictionary Version XXX.

Cohort 1 = 100μg/5mCi IV; Cohort 2 = 100μg/10mCi IV; Cohort 3 = 200μg/5mCi IV and SC.

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxxx.sas

Table 22. Vital Sign Parameters Summary Statistics Navidea Biopharmaceuticals - Study No. NAV3-24 Safety Population (N=xxx)

Page x of y

| | Vital Sign | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Group | Parameter (units) | Visit | Data Type <sup>a</sup> | Mean | Dev | n | Min | Max | Median |
| Cohort 1 IV | xxxxxxxxxx (xxx) | Pre-Injection (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | 30 min Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Cohort 2 IV | xxxxxxxxx (xxx) | Pre-Injection (Baseline) | RAW | xxx | XXX | XXX | XXX | XXX | xxx |
| | | 30 min Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Cohort 3 IV | xxxxxxxxx (xxx) | Pre-Injection (Baseline) | RAW | xxx | xxx | xxx | xxx | xxx | xxx |
| | | 30 min Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Cohort 3 SC | xxxxxxxxx (xxx) | Pre-Injection (Baseline) | RAW | xxx | xxx | xxx | xxx | xxx | xxx |
| | | 30 min Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | xxx | XXX | XXX | XXX | XXX | XXX |
| All IV Cohorts | | Dro Injection (Bacaline) | RAW | | | | | | |
| All IV Colloits | xxxxxxxxxx (xxx) | Pre-Injection (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | 30 min Post-Injection | | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

 $<sup>^{\</sup>rm a}$  RAW = data recorded in database; CFB = change from baseline Cohort 1 = 100µg/5mCi IV; Cohort 2 = 100µg/10mCi IV; Cohort 3 = 200µg/5mCi IV and SC. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 23. Vital Sign Shift Table
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

| Group | Vital Sign<br>Parameter (units) | Baseline<br>Normal/Post<br>Normal | Baseline<br>Abnormal/Post<br>Normal | Baseline<br>Normal/Post<br>Abnormal | Baseline<br>Abnormal/Post<br>Abnormal |
|---|---|---|---|---|---|
| Cohort 1 IV | xxxxxxxxx (xxx) | XXX | xxx | xxx | xxx |
| | xxxxxxxxx (xxx) | xxx | xxx | xxx | XXX |
| | xxxxxxxxx (xxx) | XXX | xxx | xxx | XXX |
| Cohort 2 IV | xxxxxxxxx (xxx) | xxx | xxx | xxx | xxx |
| | xxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | xxxxxxxxxx (xxx) | XXX | xxx | xxx | XXX |
| Cohort 3 IV | xxxxxxxxx (xxx) | XXX | xxx | xxx | xxx |
| | xxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | xxxxxxxxxx (xxx) | XXX | xxx | xxx | XXX |
| Cohort 3 SC | xxxxxxxxx (xxx) | XXX | xxx | xxx | XXX |
| | xxxxxxxxx (xxx) | xxx | XXX | xxx | XXX |
| | xxxxxxxxxx (xxx) | XXX | xxx | xxx | XXX |
| All IV Cohorts | xxxxxxxxx (xxx) | XXX | xxx | xxx | xxx |
| | xxxxxxxxxx (xxx) | xxx | XXX | XXX | XXX |
| | xxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC.

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 24. Clinical Laboratory Parameters Summary Statistics Navidea Biopharmaceuticals - Study No. NAV3-24 Safety Population (N=xxx)

| <u></u> | Laboratory Panel/ | | D | ., | Std | | | ., | |
|---|---|---|---|---|---|---|---|---|---|
| Group | Parameter (units) | Visit | Data Type <sup>a</sup> | Mean | Dev | n | Min | Max | Median |
| Cohort 1 IV | xxxxxxxxxxxx/<br>xxxxxxxxxx (xxx) | Screening (Baseline) | RAW | xxx | xxx | xxx | xxx | xxx | XXX |
| | | Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Cohort 2 IV | xxxxxxxxxxxx/<br>xxxxxxxxxx (xxx) | Screening (Baseline) | RAW | xxx | xxx | xxx | xxx | xxx | xxx |
| | | Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | xxx |
| Cohort 3 IV | Cohort 3 IV xxxxxxxxxxxx/ xxxxxxxxx (xxx) | Screening (Baseline) | RAW | xxx | xxx | xxx | xxx | xxx | xxx |
| | | Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Cohort 3 SC | xxxxxxxxxxxx/<br>xxxxxxxxxx (xxx) | Screening (Baseline) | RAW | xxx | xxx | XXX | xxx | xxx | xxx |
| | | Post-Injection | RAW | XXX | xxx | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| All IV Cohorts | xxxxxxxxxxxx/<br>xxxxxxxxxx (xxx) | Screening (Baseline) | RAW | xxx | xxx | xxx | xxx | xxx | xxx |
| | | Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | xxx |
| | | - | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

 $<sup>^</sup>a$  RAW = data recorded in database; CFB = change from baseline Cohort 1 = 100µg/5mCi IV; Cohort 2 = 100µg/10mCi IV; Cohort 3 = 200µg/5mCi IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 25. Clinical Laboratory Parameters Shift Table
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

| Group | Laboratory Panel/Parameter (units) | Baseline<br>Normal/Post<br>Normal | Baseline<br>Abnormal/Post<br>Normal | Baseline<br>Normal/Post<br>Abnormal | Baseline<br>Abnormal/Post<br>Abnormal |
|---|---|---|---|---|---|
| Cohort 1 IV | xxxxxxxxxxx/xxxxxxxx (xxx) | xxx | xxx | xxx | xxx |
| | xxxxxxxxxxxx/xxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | xxxxxxxxxxxx/xxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| Cohort 2 IV | xxxxxxxxxxx/xxxxxxxxx (xxx) | xxx | xxx | xxx | xxx |
| | xxxxxxxxxxxx/xxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | xxxxxxxxxxxx/xxxxxxxxxx (xxx) | XXX | xxx | xxx | XXX |
| Cohort 3 IV | xxxxxxxxxxx/xxxxxxxxx (xxx) | xxx | xxx | xxx | XXX |
| | xxxxxxxxxxxx/xxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | xxxxxxxxxxxx/xxxxxxxxxx (xxx) | XXX | xxx | xxx | XXX |
| Cohort 3 SC | xxxxxxxxxxxx/xxxxxxxxxx (xxx) | xxx | xxx | xxx | XXX |
| | xxxxxxxxxxxx/xxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | xxxxxxxxxxxx/xxxxxxxxxx (xxx) | XXX | xxx | xxx | XXX |
| All IV Cohorts | xxxxxxxxxxx/xxxxxxxxx (xxx) | xxx | xxx | xxx | xxx |
| | xxxxxxxxxxxx/xxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXX | XXX | XXX | XXX |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC.

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 26. Electrocardiogram Parameters Summary Statistics
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

| | | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Group | Parameter (units) | Visit | Data Typeª | Mean | Dev | n | Min | Max | Median |
| Cohort 1 IV | xxxxxxxxxxxx (xxx) | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | 30 min Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Cohort 2 IV | xxxxxxxxxxx (xxx) | Screening (Baseline) | RAW | xxx | xxx | xxx | xxx | xxx | xxx |
| COHOLC 2 IV | AAAAAAAAAAA (AAA) | 30 min Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | 30 MIN 1030 INJECTION | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFD | AAA | AAA | AAA | AAA | AAA | AAA |
| Cohort 3 IV | xxxxxxxxxxxx (xxx) | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | xxx |
| | | 30 min Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | xxx | XXX | xxx | xxx |
| Cohort 3 SC | | Caraaring (Basalina) | RAW | | | | | | |
| COHOIL 3 SC | xxxxxxxxxxxx (xxx) | Screening (Baseline) | | XXX | XXX | XXX | XXX | XXX | XXX |
| | | 30 min Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| All IV Cohorts | xxxxxxxxxxx (xxx) | Screening (Baseline) | RAW | xxx | XXX | xxx | xxx | xxx | xxx |
| | , , | 30 min Post-Injection | RAW | xxx | xxx | xxx | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | 222 | | | | | | |

a RAW = data recorded in database; CFB = change from baseline

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC.

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

## Table 27. Electrocardiogram Shift Table Navidea Biopharmaceuticals - Study No. NAV3-24 Safety Population (N=xxx)

| Group | Baseline Normal/Post<br>Normal | Baseline Abnormal/Post<br>Normal | Baseline Normal/Post<br>Abnormal | Baseline Abnormal/Post<br>Abnormal |
|---|---|---|---|---|
| Cohort 1 IV | XXX | XXX | XXX | XXX |
| Cohort 2 IV | XXX | XXX | XXX | XXX |
| Cohort 3 IV | XXX | XXX | XXX | XXX |
| Cohort 3 SC | XXX | XXX | XXX | XXX |
| All IV Cohorts | XXX | XXX | xxx | xxx |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC.

STATKING Clinical Services (month day, year)

Page x of y

Table 28. Number and Percent of Subjects Taking Concomitant Medications
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

| Medicationa: | Cohort 1<br>(N=xxx) | Cohort 2<br>(N=xxx) | Cohort 3<br>(N=xxx) | Overall<br>(N=xxx) |
|---|---|---|---|---|
| Total Number of Medications | xxx | xxx | XXX | |
| Patients Taking at Least One Medication | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| ATC Level 4 Term 1 ATC Preferred Term 1 ATC Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%) |
| ATC Level 4 Term 2 ATC Preferred Term 1 ATC Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%) |

<sup>&</sup>lt;sup>a</sup> Medications coded with WHO Coding Dictionary xxxxxxxx.

Cohort 1 = 100μg/5mCi IV; Cohort 2 = 100μg/10mCi IV; Cohort 3 = 200μg/5mCi IV and SC.

STATKING Clinical Services (month day, year)

Source Program: xxxxxxxx.sas

Page x of y

Data Listing 1. Subject Disposition Data Listing Navidea Biopharmaceuticals - Study No. NAV3-24

| | | | | Date of | |
|---|---|---|---|---|---|
| | | Subject | | Completion or | |
| | Cohort | No. | Disposition Status | Withdrawal | Withdrawal Reason |
| _ | | | | | |
| | XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXX | XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXX | XXXX | xxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxx |
| | XXXXXX | XXXX | xxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxx |
| | XXXXXX | XXXX | xxxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxx |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 2. Inclusion/Exclusion Data Listing Navidea Biopharmaceuticals - Study No. NAV3-24

| _ | Cohort | Subject | Did Subject<br>Meet All<br>Eligibility<br>Criteria? | Criterion | Criterion<br>Category | Was a<br>Waiver<br>Granted? | Is Subject<br>a Screen<br>Failure? |
|---|---|---|---|---|---|---|---|
| | XXXXXX | XXXX | XXXX | Xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX | XXXX | XXXX |
| | XXXXXX | XXXX | XXXX | Xxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX | XXXX | XXXX |
| | XXXXXX | XXXX | xxxx | Xxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX | XXXX | XXXX |
| | XXXXXX | XXXX | XXXX | Xxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX | XXXX | XXXX |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 3. Protocol Deviations Data Listing Navidea Biopharmaceuticals - Study No. NAV3-24

| | Subject | Subject | | | Deviation |
|---|---|---|---|---|---|
| Cohort | No. | Visit | Date of Deviation | Deviation Description | Category |
| XXXXXX | XXXX | XXXX | xxxxxx | xxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx |
| XXXXXX | XXXX | XXXX | xxxxxx | xxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx |
| XXXXXX | XXXX | XXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX |
| XXXXXX | XXXX | XXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 4. Demographics Data Listing Navidea Biopharmaceuticals - Study No. NAV3-24 Safety Population (N=xxx)

| | | | | | | | | | | KS |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Informed | Date | | | | | Screening | Screening | Lesions |
| | Subject | Consent | of | Age | | | | Height | Weight | at |
| Cohort | No. | Date/Time | Birth | (yrs) | Gender | Race | Ethnicity | (in) | (lb) | Screening |
| XXXXXX | XXXX | XXXXXX | XXXXXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 5. Subjects Excluded from ITD Population Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-24
All Enrolled Subjects (N=xxx)

| XXXXXX XXXX XXXXXXXXXXXXXXXXXXXXXXXXXX | XXXX |
|----------------------------------------|------|
| XXXXXX XXXX XXXXXXXXXXXXXXXXXXXXXXXXXX | XXXX |
| XXXXXX XXXX XXXXXXXXXXXXXXXXXXXXXXXXXX | XXXX |
| XXXXXX XXXX XXXXXXXXXXXXXXXXXXXXXXXXXX | XXXX |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 6. Medical History Data Listing Navidea Biopharmaceuticals - Study No. NAV3-24 Safety Population (N=xxx)

> MedDRA System Organ Class<sup>a</sup>/ MedDRA Preferred Term/

| Cohort | Subject No. | CRF Verbatim Term | Start Date | Ongoing? |
|---|---|---|---|---|
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxx | XXX |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxx | XXX |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXX | XXX |

a Medical history terms coded with MedDRA Coding Dictionary Version xxx. Cohort 1 = 100µg/5mCi IV; Cohort 2 = 100µg/10mCi IV; Cohort 3 = 200µg/5mCi IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 7. Prior and Concomitant Medications Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

WHO Drug Preferred Terma/ Verbatim Drug Name/ Indication/

| | | INGICALION/ | | | | |
|---|---|---|---|---|---|---|
| | | ATC Level 1 Code/ | Start | Stop | | |
| Cohort | Subject No. | ATC Level 4 Code | Date | Date | Route | Ongoing? |
| | | | | | | _ |
| XXXXXX | xxxxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXX | XXXXXXX | XXXXX | XXXXX |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | |
| | | xxxxxxxxxxxxxxxxxxxxxxxxx | | | | |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | |
| | | xxxxxxxxxxxxxxxxxxxxxxxxx | | | | |
| XXXXXX | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxx | XXXXXXX | XXXXX | XXXXX |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | |
| | | ******************** | | | | |

 $<sup>^{\</sup>rm a}$  Concomitant medications coded with WHO Coding Dictionary xxxxxxxxx Cohort 1 = 100µg/5mCi IV; Cohort 2 = 100µg/10mCi IV; Cohort 3 = 200µg/5mCi IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 8. Adverse Events Data Listing Navidea Biopharmaceuticals - Study No. NAV3-24 Safety Population (N=xxx)

| Cohort | Subject<br>No. | AE Start<br>Date and<br>Time/<br>End Date<br>and Time | Start Date<br>and Time of<br>most recent<br>tilmanocept<br>Injection | MedDRA System<br>Organ Classª/<br>MedDRA Preferred<br>Term/<br>CRF Verbatim Term | Treatment<br>Emergent? | Adverse<br>Drug<br>Reaction<br>(Y/N) | Severity | Relation to:<br>Tc-99m<br>tilmanocept/<br>Procedure | Serious | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxxxxx | xxxxxxx<br>xxxxxxx/<br>xxxxxxx<br>xxxxxxx | xxxxxx | ************************************** | xxx | xxx | xxxxxxx | xxxxxxx/<br>xxxxxxxx | xxx | xxxxxx<br>x |
| xxxxxx | xxxxxxxx | xxxxxxx<br>xxxxxxx/<br>xxxxxxx<br>xxxxxx | xxxxxx | ************************************** | xxx | xxx | xxxxxxx | xxxxxxx/<br>xxxxxxxx | xxx | xxxxxx<br>x |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version xxx.

Cohort 1 = 100μg/5mCi IV; Cohort 2 = 100μg/10mCi IV; Cohort 3 = 200μg/5mCi IV and SC.

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxxx.sas

Page x of y

Data Listing 9. Subject Laboratory Profiles - Hematology Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

| Normal | Range |
|--------|-------|
|--------|-------|

| Cohort | Subject<br>No. | Visit | Sample Date/<br>Time | Parameter (Unit: | s) Result | Lab Low | Lab High | Clin.<br>Sig? |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxx | xxxxxxx<br>xx:xx | xxxxxxxxxxx (xx | x) xxx | xxx | xxx | xxx |
| | | | | xxxxxxxxxxx (xx | x) xxx | xxx | XXX | XXX |
| | | | | xxxxxxxxxxxx (xx | x) xxx | XXX | XXX | XXX |
| | | | | xxxxxxxxxxx (xx | x) xxx | XXX | XXX | XXX |
| | | | | xxxxxxxxxxx (xx | x) xxx | XXX | XXX | XXX |
| | | | | xxxxxxxxxxx (xx | x) xxx | XXX | XXX | XXX |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 10. Subject Laboratory Profiles - Serum Chemistry Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

Normal Range

| Cohort | Subject<br>No. | Visit | Sample Date/<br>Time | Parameter (U | nits) | Result | Lab Low | Lab High | Clin.<br>Sig? |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxx<br>xx:xx | xxxxxxxxxx | (xxx) | xxx | xxx | xxx | xxx |
| | | | | xxxxxxxxxxx | (xxx) | XXX | XXX | XXX | xxx |
| | | | | XXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 11. Subject Laboratory Profiles - Urinalysis Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

## Normal Range

| Cohort | Subject<br>No. | Visit | Sample Date/<br>Time | Parameter (U | Jnits) | Result | Lab Low | Lab High | Clin.<br>Sig? |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxx | xxxxxxx<br>xx:xx | xxxxxxxxxx | (xxx) | xxx | xxx | xxx | xxx |
| | | | ***** | xxxxxxxxxxx | (xxx) | xxx | xxx | xxx | xxx |
| | | | | xxxxxxxxxxx | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |
| | | | | XXXXXXXXXXX | (xxx) | XXX | XXX | XXX | XXX |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC.

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

## Data Listing 12. Electrocardiogram Data Listing Navidea Biopharmaceuticals - Study No. NAV3-24 Safety Population (N=xxx)

| | ECG Assessment,<br>Abnormal, Spec | QTcF<br>Interval<br>(msec) | QT<br>Interval<br>(msec) | QRS<br>Duration<br>(msec) | PR<br>Interval<br>(msec) | Heart<br>Rate<br>(bpm) | Time | Date | Visit | Subject<br>No. | Cohort |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ĸ/ | xxxxxxx/ | xxxxx | xxxxx | xxxxx | xxxxx | xxxxx | xxxxx | xxxxx | xxxxxxx | xxxx | xxxxxx |
| | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx/ | xxxxx | xxxxx | xxxxx | xxxxx | xxxxx | xxxxx | xxxxx | xxxxxx | | |
| XXXXXX | XXXXXXXXXXXXXXXXX | | | | | | | | | | |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 13. Physical Exam Data Listing Navidea Biopharmaceuticals - Study No. NAV3-24 Safety Population (N=xxx)

| | Subject | | | | | |
|---|---|---|---|---|---|---|
| Cohort | No. | Visit | Date | Body System | Result | Abnormality |
| XXXXXX | XXXX | XXXXXXX | XXXXXXX | General Appearance | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | | Skin | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Eyes, Ears, Nose, Throat | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Head and Neck | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Heart | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Lungs | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Abdomen | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Lymph Nodes | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Musculoskeletal | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | CNS/Neurological | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 14. Vital Signs Data Listing Navidea Biopharmaceuticals - Study No. NAV3-24 Safety Population (N=xxx)

| | | | | | | Systoli | c Blood | Diastol | ic Blood | Heart | Rate | Respi | rations |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Temperat | ture (°F) | Pressur | e (mmHg) | Pressur | e (mmHg) | (bj | om) | per N | Minute |
| | Subject | Visit/ | | | Normal | | Normal | | Normal | | Normal | | Normal |
| Cohort | No. | Date | Time | Value | (Y/N) | Value | (Y/N) | Value | (Y/N) | Value | (Y/N) | Value | (Y/N) |
| xxxxxx | xxxx | xxxxxxx/<br>xxxxxx | xxxxx | xxx | Х | xxx | х | xxx | х | xxx | Х | xxx | х |
| | | | xxxxx | xxx<br>xxx | x<br>x | xxx<br>xxx | X<br>X | xxx<br>xxx | x<br>x | xxx<br>xxx | x<br>x | xxx<br>xxx | x<br>x |
| xxxxxx | xxxx | xxxxxxx/<br>xxxxxx | xxxxx | XXX | х | XXX | Х | xxx | Х | xxx | х | xxx | Х |
| | | | XXXXX | XXX | X | XXX | X | XXX | X | XXX | X | XXX | X |
| | | | XXXXX | XXX | X | XXX | X | XXX | X | XXX | X | XXX | X |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 15. Study Drug Administration Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

| | Subject | Date/<br>Time of | Anatomic<br>Location<br>of | Pre-Injection<br>Radioactivity<br>(mCi)/Time of | Post-<br>Injection<br>Radioactivity<br>(mCi)/Time of | Calculated Amount of Administered Radioactivity | Calculated<br>Mass Dose | Lot |
|---|---|---|---|---|---|---|---|---|
| Cohort | No. | Injection | Injection | Measurement | Measurement | (mCi) | (µg) | Number |
| xxxxxx | xxxx | xxxxxxxx/<br>xxxx | xxxxxxx | xxx/<br>xxxx | xxx/<br>xxxx | xxx | xxx | XXX |
| xxxxxx | xxxx | xxxxxxxx/<br>xxxx | xxxxxxx | xxx/<br>xxxx | xxx/<br>xxxx | xxx | xxx | xxx |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 16. Post-Injection Imaging Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-24
ITD Population (N=xxx)

| | | | Start | |
|--------|---------|---------|---------|---------------|
| | | | Time of | SPECT/CT |
| | Subject | Date of | Planar | Imaging Start |
| Cohort | No. | Imaging | Imaging | Time |
| XXXXXX | XXXX | XXXXXX | xx:xx | xx:xx |
| XXXXXX | XXXX | XXXXXX | XX:XX | xx:xx |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 17. Quantitative Imaging Results Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-24

ITD Population (N=xxx)

| | Cohort | Subject<br>No. | Identified Clinically or with Imaging? | Lesion <sup>a</sup> | Average<br>Pixel<br>Intensity | Average<br>Background<br>Intensity | Percent Above<br>Background |
|---|---|---|---|---|---|---|---|
| • | xxxxxx | xxxx | xxxxxx | xxxxxxxxx | xxxx | xxxx | xxxx |
| | XXXXXX | XXXX | xxxxxxx | xxxxxxxxx | XXXX | xxxx | xxxx |

 $<sup>^{\</sup>rm a}$  Lesions previously identified clinically and biopsied. Cohort 1 = 100µg/5mCi IV; Cohort 2 = 100µg/10mCi IV; Cohort 3 = 200µg/5mCi IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 18. Qualitative Imaging Results Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-24
ITD Population (N=xxx)

| Cohort | Subject<br>No. | Identified Clinically or with Imaging? | Lesion <sup>a</sup> | Reader<br>Visualization |
|---|---|---|---|---|
| XXXXXX | xxxx | xxxxxx | xxxxxxxxx<br>xxxxxxxxx | XXX<br>XXX |

 $<sup>^{\</sup>rm a}$  Lesions previously identified clinically and those additional lesions identified on imaging. Cohort 1 = 100µg/5mCi IV; Cohort 2 = 100µg/10mCi IV; Cohort 3 = 200µg/5mCi IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 19. Lesion Biopsy Results Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-24

ITD Population (N=xxx)

| Cohort | Subject<br>No. | Biopsy<br>Date/Time | Location of<br>Lesion <sup>a</sup> | Measurement<br>of Biopsy<br>(mm) | HHV8<br>RFU | Proportion<br>of CD206-<br>expressing<br>Cells | Proportion of<br>HHV8-<br>expressing<br>Cells |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxxx / | xxxxxxxxx | xxx | xxxxx | xxxx | xxxx |
| xxxxxx | xxxx | xx:xx<br>xxxxxxxxxx /<br>xx:xx | xxxxxxxx | xxx | xxxxx | xxxx | xxxx |

 $<sup>^{\</sup>rm a}$  Lesions previously identified clinically and biopsied. Cohort 1 = 100µg/5mCi IV; Cohort 2 = 100µg/10mCi IV; Cohort 3 = 200µg/5mCi IV and SC. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 20. Clinical KS Lesion Assessment Listing Navidea Biopharmaceuticals - Study No. NAV3-24 ITD Population (N=xxx) Part 1 of 2

| Cohort <sup>a</sup> | Subject<br>No. | Assessment<br>Date | KS<br>Diagnosis<br>Date | Biopsy<br>Confirmation<br>Date | KS<br>Classification <sup>b</sup> |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxxx | xxxx | xxxx | x |
| XXXXXX | XXXX | XXXXXXXXX | XXXX | xxxx | x |

 $<sup>^{\</sup>rm a}$  Cohort 1 = 100 $\mu$ g/5mCi IV; Cohort 2 = 100 $\mu$ g/10mCi IV; Cohort 3 = 200 $\mu$ g/5mCi IV and SC.

b 1 = Confirmed cutaneous or oral lesions without edema, 2 = Confirmed cutaneous or oral lesions with edema, 3 = Confirmed cutaneous or oral lesions with or without edema and suspected or confirmed non-cutaneous lesions. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 20. Clinical KS Lesion Assessment Listing
Navidea Biopharmaceuticals - Study No. NAV3-24

ITD Population (N=xxx)

Part 2 of 2

| Suspected Non- Cutaneous KS/Location Symptomology | Confirmed Non- Cutaneous KS/Location Symptomology | Number<br>of<br>Overall<br>Lesions | Lesion<br>Number | Lesion<br>Type/Location | Edema Present?/<br>Edema Scale |
|---|---|---|---|---|---|
| xxxx | х | XXX | XX<br>XX | xxxx/xxxxx<br>xxxx/xxxxx | xxx/x<br>xxx/x |
| xxxx | х | xxx | xx<br>xx<br>xx | xxxx/xxxxx<br>xxx/xxxx<br>xxxx/xxxxx | xxx/x<br>xxx/x<br>xxx/x |

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Data Listing 21. Telephone Follow Up Contact Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-24
Safety Population (N=xxx)

| Cohort | Was Telephone Subject Contact hort No. Performed? | | Date of Contact | Time of<br>Contact | Any AEs Since<br>Previous Visit? | Changes in Medications<br>Since Previous Visit? |
|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxx | xxxx | xxxx | xxxx | xxxx |
| xxxxxx | xxxx | xxxx | xxxx | xxxx | xxxx | xxxx |

Cohort 1 =  $100\mu g/5mCi$  IV; Cohort 2 =  $100\mu g/10mCi$  IV; Cohort 3 =  $200\mu g/5mCi$  IV and SC. STATKING Clinical Services (DD-MMM-YYYY)